CLINICAL TRIAL: NCT03419624
Title: A 28-week, Multi-center Randomized, Double-blind, Placebo-controlled Study to Evaluate the Potential of Dapagliflozin Plus Exenatide in Combination With High-dose Intensive Insulin Therapy Compared to Placebo in Obese Insulin-resistant Patients With Type 2 Diabetes Mellitus (Proof-of-concept Study)
Brief Title: The Potential of Dapagliflozin Plus Exenatide in Obese Insulin-resistant Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Delay in patient enrolment
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKE-DapEx-001
Record Dates: First submitted 2018-01-17; First posted 2018-02-05 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
Keywords: Dapagliflozin; Exenatide; high-dose insulin therapy; SGLT-2 inhibitor; GLP-1 receptor agonist
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Exenatide; Insulin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapagliflozin plus Exenatide (Experimental): Dapagliflozin (10mg orally once daily) plus Exenatide (2mg subcutaneous once-weekly injection) as add-on to high-dose intensive insulin therapy
  Interventions: Drug: Dapagliflozin 10mg; Drug: Exenatide 2 mg [Bydureon]; Drug: Insulin; Drug: Metformin, if taken before
- Placebo plus Placebo (Placebo Comparator): Placebo (film-coated tablet once daily) plus Placebo (subcutaneous once-weekly injection) as add-on to high-dose intensive insulin therapy
  Interventions: Drug: Placebo Oral Tablet; Drug: Placebo injection; Drug: Insulin; Drug: Metformin, if taken before
- Placebo plus Exenatide (Active Comparator): Placebo (film-coated tablet once daily) plus Exenatide (2mg subcutaneous once- weekly injection) as add-on to high dose intensive insulin therapy
  Interventions: Drug: Exenatide 2 mg [Bydureon]; Drug: Placebo Oral Tablet; Drug: Insulin; Drug: Metformin, if taken before

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin 10 mg tablet once daily
  Arms: Dapagliflozin plus Exenatide
Drug: Exenatide 2 mg [Bydureon] — Exenatide 2 mg injection once weekly
  Arms: Dapagliflozin plus Exenatide; Placebo plus Exenatide
Drug: Placebo Oral Tablet — Placebo oral tablet once daily
  Arms: Placebo plus Exenatide; Placebo plus Placebo
Drug: Placebo injection — Placebo injection once weekly
  Arms: Placebo plus Placebo
Drug: Insulin — daily Insulin injections
Drug: Metformin, if taken before — If the Patient has taken Metformin prior to enrollment, he or she will continue to take it.

SUMMARY:
This is a 28-week, multi-center, randomized, double-blind, placebo-controlled trial to study a potential synergistic effect of Dapagliflozin plus Exenatide once-weekly in combination with high-dose intensive insulin therapy compared to Placebo in obese insulin-resistant patients with Type 2 Diabetes mellitus (T2DM) and inadequate glycemic control (HbA1c≥8.0% and ≤ 11.0%).

DETAILED DESCRIPTION:
In this proof-of-concept study the potential of treatment with Dapagliflozin plus Exenatide added to high-dose intensive insulin therapy compared to Placebo added to high-dose intensive insulin with active insulin up-titration for change in HbA1c from baseline to week 28 shall be explored and generate initial data on the primary outcome. We hypothesize that SGLT-2 inhibition and GLP-1 receptor agonism may be a rational combination therapy that addresses a broad range of pathophysiological defects associated with T2DM in obesity and may reduce HbA1c levels in patients with severe insulin resistance. In a third treatment arm, patients will be treated with Exenatide monotherapy added to high-dose intensive Insulin therapy to study additive effects of Dapagliflozin and Exenatide.

ELIGIBILITY:
For inclusion in the study patients should fulfill the following key criteria:

1. Informed Consent can be obtained prior to any study procedures.
2. Patient is able to read, understand and sign the Informed Consent.
3. HbA1c ≥ 8.0% and ≤ 11.0% based on laboratory results
4. Currently treated with a stable TDID ≥ 80 U at least 3 months prior to enrolment
5. Patients who are receiving metformin must be on a stable total daily dose ≥ 1500 mg or the maximum tolerated dose of metformin within 3 months prior to enrolment
6. BMI of ≥ 30 kg/m2 at enrolment
7. Male or female and ≥18 and ≤75 years old at time of informed consent
8. For female patients:

   * Not breastfeeding.
   * Negative pregnancy test result (human chorionic gonadotropin, beta subunit [βhCG]) at Visit 0 (Screening) and Visit 1 (randomization) -not applicable to hysterectomized and post-menopausal females.
   * If of childbearing potential (including perimenopausal women who have had a menstrual period within 1 year), must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, ie, less than 1% per year, when used consistently and correctly, such as implants, injectables, hormonal contraceptives [pills, vaginal rings, or patches], some intrauterine contraceptive devices [levonorgestrel-releasing or copper-T], tubal ligation or occlusion, or a vasectomized partner) during the entire duration of the study. As applicable, all methods must be in effect prior to receiving the first dose of study medication.
   * Must practice appropriate birth control as stated above for 10 weeks after the last dose of study medication.
9. Patients who are receiving the following medications must be on a stable treatment regimen for a minimum of 2 months prior to Visit 0 (Screening):

   * Antihypertensive agents
   * Thyroid replacement therapy
   * Antidepressant agents

Exclusion Criteria:

1. Diagnosis of Type 1 Diabetes
2. History of diabetic ketoacidosis, hyperosmolar coma or corticosteroid-induced Type 2 diabetes
3. Patients with significant thyroid disease
4. Patients with history of acute or chronic pancreatitis
5. Clinically significant cardiovascular disease or procedure within 3 months prior to enrolment or expected to require coronary revascularization procedure
6. Presence of history of severe congestive heart failure (NYHA III and IV)
7. Creatinin-Clearance of < 60 ml/min based on local laboratory results
8. Concomitant medication with loop diuretics
9. Patients who, as judged by the investigator, may be at risk for dehydration or volume depletion that may affect the patient's safety (including e.g. patients with a history of Diabetes insipidus)
10. Pregnant women
11. Administration of any other antidiabetic therapy, other than insulin (see inclusion criterion no.4 and 5) and metformin with a stable total daily dose ≥ 1500 mg or the maximum tolerated dose of metformin within 3 months prior to enrolment
12. History of, or currently have, acute or chronic pancreatitis, or have triglyceride concentrations ≥ 700 mg/dL (≥ 7.98 mmol/L) at Visit 0 (Screening).
13. History or presence of inflammatory bowel disease or other severe GI diseases, particularly those which may impact gastric emptying, such as gastroparesis or pyloric stenosis.
14. History of gastric bypass surgery or gastric banding surgery, or either procedure is planned during the time period of the study. Current use of gastric balloons is also excluded.
15. Significant hepatic disease, including, but not limited to, acute hepatitis, chronic active hepatitis, or severe hepatic insufficiency, including patients with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or total bilirubin (TB) >2 mg/dL (>34.2 μmol/L) (patients with TB >2 mg/dL [>34.2 μmol/L] and documented Gilbert's syndrome will be allowed to participate).
16. Known history of hepatotoxicity with any medication
17. Known history of severe hepatobiliary disease.
18. Positive serological test for hepatitis B or hepatitis C.
19. Known or suspected human immunodeficiency virus (HIV) infection.
20. History of organ transplantation.
21. Presence or history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2 (MEN 2) OR a family history of medullary thyroid carcinoma or MEN 2.
22. Malignancy (with the exception of basal and squamous cell carcinoma of the skin) within 5 years of Visit 0 (Screening).
23. Hemoglobinopathy, hemolytic anemia, or chronic anemia (haemoglobin concentration <11.5 g/dL [115 g/L] for males, <10.5 g/dL [105 g/L] for females) or any other condition known to interfere with the HbA1c methodology.
24. Patients with abnormal test results of hematocrit (hematocrit > 50% for men; hematocrit > 47% for women)
25. Has donated blood or had a significant blood loss within 2 months of first dose of study medication or is planning to donate blood during the study.
26. Has donated plasma within 7 days prior to first dose of study medication.
27. Any exposure to Exenatide (including BYETTA®, BYDUREON, or exenatide suspension).
28. Any exposure to Dapagliflozin or any SGLT-2 inhibitor.
29. Has been treated, is currently being treated, or is expected to require or undergo treatment with any of the following treatment excluded medications:

    * Any DPP-4 inhibitor within 3 months prior to Visit 0 (Screening).
    * Any GLP-1 analog within 1 year prior to Visit 0 (Screening).
    * Systemic corticosteroids within 3 months prior to Visit 0 (Screening) by oral, intravenous, intra-articular, or intramuscular route; or potent, inhaled, or intrapulmonary (including ADVAIR) steroids known to have a high rate of systemic absorption. For examples of excluded steroids, refer to Section 7.7.
    * Prescription or over-the-counter weight loss medications within 3 months prior to Visit 0 (Screening).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from baseline (week 0) to week 28 | 28 weeks
  To compare the absolute change from baseline in HbA1c at week 28 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy

SECONDARY OUTCOMES:
Change in HbA1c from baseline (week 0) to week 14 | 14 weeks
  To compare the absolute change in HbA1c from baseline at week 0 to week 14 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy
Change in total body weight from baseline (week 0) to week 14 and 28 | 28 weeks
  To compare the change in total body weight from baseline at week 0 to week 14 and 28 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy
Change in BMI from baseline (week 0) to week 14 and 28 | 28 weeks
  To compare the change in BMI from baseline at week 0 to week 14 and 28 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy
Change in FPG from baseline (week 0) to week 14 and 28 | 28 weeks
  To compare the change in fasting plasma glucose (FPG) from baseline at week 0 to week 14 and 28 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy
Change in TDID from baseline (week 0) to week 14 and 28 | 28 weeks
  To compare the change in total daily insulin dose (TDID) from baseline at week 0 to week 14 and 28 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy
Proportion of patients achieving HbA1c of ≤ 7% at week 28 compared to baseline | 28 weeks
  To compare the number of patients achieving HbA1c of ≤ 7% at week 28 compared to baseline at week 0 between Dapagliflozin plus Exenatide, Placebo or Exenatide monotherapy added to high-dose intensive insulin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jens Aberle, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (4):
- Germany (4):
  - Diabeteszentrum Oldenburg, Oldenburg, Lower Saxony
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Diabetologische Schwerpunktpraxis Harburg, Hamburg
  - Gemeinschaftspraxis für Innere Medizin und Diabetologie, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prasad-Reddy L, Isaacs D. A clinical review of GLP-1 receptor agonists: efficacy and safety in diabetes and beyond. Drugs Context. 2015 Jul 9;4:212283. doi: 10.7573/dic.212283. eCollection 2015. PMID 26213556
- [Background] Wilding JP, Woo V, Soler NG, Pahor A, Sugg J, Rohwedder K, Parikh S; Dapagliflozin 006 Study Group. Long-term efficacy of dapagliflozin in patients with type 2 diabetes mellitus receiving high doses of insulin: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):405-15. doi: 10.7326/0003-4819-156-6-201203200-00003. PMID 22431673
- [Background] Finkelstein EA, Khavjou OA, Thompson H, Trogdon JG, Pan L, Sherry B, Dietz W. Obesity and severe obesity forecasts through 2030. Am J Prev Med. 2012 Jun;42(6):563-70. doi: 10.1016/j.amepre.2011.10.026. PMID 22608371
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR. Management of hyperglycaemia in type 2 diabetes: a patient-centered approach. Position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2012 Jun;55(6):1577-96. doi: 10.1007/s00125-012-2534-0. Epub 2012 Apr 20. No abstract available. PMID 22526604
- [Background] Tatarkiewicz K, Polizzi C, Villescaz C, D'Souza LJ, Wang Y, Janssen S, Parkes DG. Combined antidiabetic benefits of exenatide and dapagliflozin in diabetic mice. Diabetes Obes Metab. 2014 Apr;16(4):376-80. doi: 10.1111/dom.12237. Epub 2013 Dec 9. PMID 24251534
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B. Management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: update regarding thiazolidinediones: a consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2008 Jan;31(1):173-5. doi: 10.2337/dc08-9016. No abstract available. PMID 18165348
- [Background] Wangnoo SK, Sethi B, Sahay RK, John M, Ghosal S, Sharma SK. Treat-to-target trials in diabetes. Indian J Endocrinol Metab. 2014 Mar;18(2):166-74. doi: 10.4103/2230-8210.129106. PMID 24741511
- [Background] Holman R. Metformin as first choice in oral diabetes treatment: the UKPDS experience. Journ Annu Diabetol Hotel Dieu. 2007:13-20. PMID 18613325
- [Background] Blevins T, Pullman J, Malloy J, Yan P, Taylor K, Schulteis C, Trautmann M, Porter L. DURATION-5: exenatide once weekly resulted in greater improvements in glycemic control compared with exenatide twice daily in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011 May;96(5):1301-10. doi: 10.1210/jc.2010-2081. Epub 2011 Feb 9. PMID 21307137
- [Background] Diamant M, Van Gaal L, Stranks S, Northrup J, Cao D, Taylor K, Trautmann M. Once weekly exenatide compared with insulin glargine titrated to target in patients with type 2 diabetes (DURATION-3): an open-label randomised trial. Lancet. 2010 Jun 26;375(9733):2234-43. doi: 10.1016/S0140-6736(10)60406-0. PMID 20609969
- [Background] Sharma S, Jain S. Prevalence of Obesity among Type-2 Diabetics. J Hum Ecol 2009;25:31-5.
- [Background] Dixon JB, O'Brien PE. Health outcomes of severely obese type 2 diabetic subjects 1 year after laparoscopic adjustable gastric banding. Diabetes Care. 2002 Feb;25(2):358-63. doi: 10.2337/diacare.25.2.358. PMID 11815510
- [Background] 2012. Guideline on clinical investigation of medicinal products in the treatment or prevention of diabetes mellitus n.d. ema.europa.eu.
- [Background] Anderson SL. Dapagliflozin efficacy and safety: a perspective review. Ther Adv Drug Saf. 2014 Dec;5(6):242-54. doi: 10.1177/2042098614551938. PMID 25436106
- [Background] EMA confirms recommendations to minimise ketoacidosis risk with SGLT2 inhibitors for diabetes 2016. www.ema.europe.eu.
- [Background] Frias JP, Guja C, Hardy E, Ahmed A, Dong F, Ohman P, Jabbour SA. Exenatide once weekly plus dapagliflozin once daily versus exenatide or dapagliflozin alone in patients with type 2 diabetes inadequately controlled with metformin monotherapy (DURATION-8): a 28 week, multicentre, double-blind, phase 3, randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Dec;4(12):1004-1016. doi: 10.1016/S2213-8587(16)30267-4. Epub 2016 Sep 16. PMID 27651331
- [Background] FDA approves Farxiga to treat type 2 diabetes. 2014 n.d. fda.gov.
- [Background] FDA Approves Bydureon Pen. 2014 n.d. drugs.com.